CLINICAL TRIAL: NCT04696107
Title: Effectiveness of Coping Strategies on the Control of Musculoskeletal Chronic Non-Cancer Pain and Quality of Life: A Randomized Clinical Trial
Brief Title: Effectiveness of Coping Strategies on the Control of Chronic Non-Cancer Pain and Quality of Life (CNCP_CopQol)
Acronym: CNCP_CopQol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital San Juan de Dios del Aljarafe de Sevilla (Other)
Collaborators: University of Seville (Other); Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSJDA-20.1
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain; Musculoskeletal Diseases; Quality of Life; Pain Measurement
Keywords: Chronic Non-Cancer Pain; Quality of life; Pain control; Coping; Patient education; Psychoeducative intervention
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Diseases; Agnosia

STUDY DESIGN:
Intervention Model Description: A triple blinded, Randomized, Parallel-Group Clinical Trial.
  1. Patients who meet the inclusion criteria are informed, voluntarily agree to participate and give signed consent at their Primary Care Center, will be included in the study. In the Investigation Unit of the Hospital San Juan De Dios del Aljarafe they will be anonymised using a table where their medical history number will be assigned an order number, which will serve as identification. They will also be randomized by permuted blocks.
  2. Telephone surveys: A professional of the Hospital San Juan de Dios del Aljarafe will be responsible for taking all questionnaires by telephone at the beginning, per month, three months and six months of inclusion for each patient.
  3. Psychoeducational intervention: The two professionals who teach the workshops are hospital workers with training in Pain Neuroscience and Coaching.
  4. Data analysis: by a biostatistics expert. No professional can access the rest of the information of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: After randomization and assignment to each arm, the masking will be triple ( researcher, evaluator of results, participant):
  * Researchers: All the professionals who participate in the study will only do so in a single specific stage and will be blinded to the assignment and development of others.
  * Evaluators of results: The results will be analyzed by an independent statistical professional and the evaluation of the response will be carried out by researchers who do not know the group to which each patient belongs.
  * Participant: Patients will be blinded for up to six months of follow-up. Then they will know the group to which they belong and will be invited to do the workshop if they have belonged to the control group.
  We don't believe that it is possible that a patient emergency unmasking will be required due to secondary effects, even so, the Patient Safety Committee will inform of any incident.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Standard pharmacological treatment aimed at controlling mCNCP with four-week face to face psychoeducational intervention.
  Interventions: Behavioral: Psychoeducative intervention
- Control Group (No Intervention): Standard pharmacological treatment aimed at controlling mCNCP without psychoeducational intervention.

INTERVENTIONS:
Behavioral: Psychoeducative intervention — This workshop is centred in psychoeducational and training action in emotional self-regulation in a group modality and participatory character, aimed at patients with mCNCP to acquire basic knowledge in:
  * Neurology and psychoneuroimmunology.
  * The role of beliefs in our manifestation of the disease.
  * Body language and modulation of pain perception.
  * Relaxation body-mind techniques.
  * Creative visualization for pain management.
  * Mirror feed-back.
  The workshop will take place at the Hospital San Juan de Dios del Aljarafe, in four weeks, once a week, three hours each. Until now, the attendance was 24 patients per workshop. After the pandemic, we will reduce to 15 to increase safety distance. We will also conduct a telephone survey of each patient on symptoms of Covid infection in the 24 hours prior to the workshop.
  Arms: Intervention Group

SUMMARY:
* Introduction and objectives: Non-pharmacological interventions in patients with musculoskeletal chronic non-cancer pain (mCNCP) are positioning themselves as an essential pillar in treatment along with pharmacological and interventional treatment. Training the patient in psycho-educational interventions focused on the neuroscience of pain and accompanying them towards a better coping of their disease can decrease the perception of pain and improve their quality of life. A previous pilot study, developed by the researchers about this type of interventions, identified as relevant data an improvement in the quality of life (QoL) of patients with mCNCP with a significant decrease in pharmacological consumption, and a high degree of satisfaction on the part of the user through the analysis of PROMs (patient-reported outcome measures). The main objective of this study is to know the effectiveness in the perception of pain through the Verbal Numerical Rating Scale (VNRS) and in the quality of life through the EuroQol-5D (EQ-5D) questionnaire of a psychoeducational intervention focused on emotional coping strategies, in patients with mCNCP in the Primary Care Centres of Public Health System of Aljarafe-Sevilla Norte Area (Spain). Secondarily, the consumption of health resources associated with mCNCP, the adherence to treatment, the influence of social, emotional, and family variables will be studied by the researchers in the two groups of patients on each telephone assessment.
* Methodology: Prospective, randomized, triple-blind (patient, investigator, and analysis) and controlled clinical trial. Participants with mCNCP in follow-up in Primary Care without clinical control with the treatment scheduled and who agree to participate in the study will be randomized by blocks permuted to receive treatments and standard care (control group) or these same care plus a psychoeducational intervention (experimental group). This intervention consists of an emotional self-regulation training program of four face-to-face sessions of 3 hours each, over a four-week period. The study will include 144 participants (72 for each arm). Patient follow-up will be telephone at the time of inclusion, at month, three, and six months. A descriptive and multivariate analysis will be done with the patients' research data associated with pain or QoL, post-intervention.
* Ethics and dissemination: The study will be carried out following the Helsinki Declaration and is approved by the Committee on Ethics of Research of Virgen Macarena- Virgen del Rocío university hospitals in Seville, Spain (code 1589-N-19). The results of the trial will be published under CONSORT regulations and SPIRIT guideline.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE

   Many people with mCNCP experience stress, fear and depression. These emotions, mental states and their associated behaviours often act as aggravating factors, amplifying the perception of pain (1-3). As a result, the same stimulus produces more suffering and begins a vicious circle. In this context, the acceptance and engagement therapy (ACT) and mindfulness-based stress reduction (MBSR) can be very helpful in managing chronic pain. These practices allow the patients to focus on participating in valuable activities and finding personally relevant objectives, improving their coping in this situation.

   Based on systematic reviews the investigators can confirm that body-mind therapies, especially MBSR and pain neuroscience education show benefits in a different kind of noncancer chronic pain in the adult such as reducing the severity of pain and functional limitation, maintaining the positive effects in the long term. On the other hand, related to a growing interest in reducing the use of opioid medications, it is also important to determine if one of the results of psychological approaches is the decrease in drug use, and as a consequence, a decrease in health cost per patient. Although this is one of the benefits assumed, studies about the association between pain management or self-control interventions and dependence on painkillers are lacking. There are not enough data about the behavioral intervention effects on the use of pain medication but initially points to a reduction. Therefore, it is necessary to focus on the management of the mCNCP integrally, incorporating non-pharmacological therapies that provide the patients with skills to face the illness and, above all, empower themselves through information and training the self-care.

   Researchers propose this clinical trial to demonstrate the effectiveness of a psychoeducational intervention focused on emotional coping in the control of symptoms, QoL and consumption of analgesics and health resources in patients with mCNCP.
2. RESEARCH QUESTION

   The early and integratively detection and approach of mCNCP are the main tools to decrease its prevalence and negative effects on both the patient life and the Health System. Scientific evidence supports body-mind therapies and patient education in pain neuroscience that enable a positive adaptive response that appears to improve functionality and QoL in people affected by mCNCP. That is why the research question directed by this investigation is: "Can a psychoeducational intervention focused on emotional coping reduce the pain perception and improve the QoL of adult patients with mCNCP treated in Public Primary Health Centre of the Aljarafe-North Seville Area?"
3. OBJECTIVES:

   3.1. Main objective: Know the effectiveness in pain perception through VNRS and QoL through the EQ-5D scale of psychoeducational intervention focused on emotional coping strategies, in participants with mCNCP in the Public Health Centers of the Aljarafe-North Seville Area.

   3.2. Specific objectives:
   * Identify the sociodemographic, clinical, psychological, and functional characteristics of mCNCP patients based on disease type and sex.
   * Compare scores on pain perception and QoL between the workshop group and the control group before the intervention and throughout follow-up.
   * Evaluate changes in analgesic pharmacological consumption in conventionally treated participants versus those who also receive psychoeducational intervention focused on emotional coping and self-control techniques.
   * Analyse the frequentation of health services and the number of days of work disability caused by the intensification of pain in conventionally treated patients compared to those receiving the psychoeducational intervention.
   * Assess the influence of global family functioning and emotional coping on the experience of pain through the Family Apgar Scale and the Reduced Chronic Pain Coping Questionnaire, respectively.
   * Assess the impact of the intervention on sleep quality and co-existing sleep disorders.
   * Detect predictors of the effectiveness of psychoeducational intervention focused on emotional coping and identify profiles of patients more sensitive to modify the pain perception or quality of life through psychoeducational intervention.
4. SAMPLE SIZE

   Based on a previous pilot study and accepting an alpha risk of 0.05 and a beta risk of 0.2 in a bilateral contrast, 72 subjects are required in the first group and 72 in the second to detect a difference equal to or greater than 0.07 on 1 on the EQ-5D scale between the two groups. The common standard desviation is assumed to be 0.16 and a correlation coefficient between the initial and final measurement of 0.61. A loss to follow-up rate of 10% has been estimated. (Total = 144).
5. RECRUITMENT

   Participants will be recruited for clinical trials at Primary Care Centres of Public Health System of Spain through the identification in the Chronic Non-Cancer Pain patient registry (database).
6. ASSIGNMENT OF INTERVENTION. SEQUENCE GENERATION Participants will be randomly assigned to a control or experimental group by permutations of two elements (the number of groups) taken four by four (the size of the block): AABB, ABAB, ABBA, BAAB, BABA and BBAA. Finally, the blocks are randomly ordered from one to six and the participants are successively assigned to the corresponding option, completing the blocks in the order established at random. In this way, with every four participants assigned the size of the two groups will be equalized.
7. DATA MANAGEMENT

   In this clinical trial, all data will be entered electronically except for comments made by participants at the end of each workshop in the intervention group. Participant data will be stored in numerical order in a secure location accessible only to professionals who enter and analyze the data. Participant files will be kept for a period of 3 years after completion of the study.
8. STATISTICAL ANALYSIS

   First, a descriptive analysis of all the variables will be carried out. Qualitative variables will be presented by absolute and relative frequencies and quantitative variables by the mean and standard deviation or median and interquartile range, depending on whether or not a normal distribution is followed.

   In the second stage, an intention-to-treat analysis will be developed. To perform the analysis between different variables or factors that could influence the results, the Chi-square test or Fisher's exact test will be used for qualitative variables and the Student's t-test and ANOVA or U of Mann Whitney and Kruskal Wallis for quantitative variables, depending on whether a normal distribution is followed. To explore the relationship between the dependent variables and the participants sociodemographic, psychosocial and clinical characteristics, the appropriate tests will be used in each situation (Student's T-test, ANOVA, Pearson's correlation coefficient) or the non-parametric alternatives if necessary (U of Correlation of Mann Whitney, Kruskal Wallis and Spearman). For the comparative analysis between the two intervention groups and in the repeated samples of each patient, contrast tests will be used for independent and related samples, respectively.

   To control the possible confounding effect of some variables and/or the possible interactions on the global score of EQ-5D and VNRS, multivariate regression models will be run, taking into account the linear or non-linear relationship of the possible predictors with the outcomes. The analyzes will also be carried out with relevant study strata such as the patient's profile, detected from the cluster analysis, according to variables associated with the characteristics of pain and its etiopathogenesis.

   The level of statistical significance will be set at p less than 0.05. The statistical analysis will be carried out with the SPSS package, version 19.0. and R Studio.
9. COMMITTEES

   - Principal Investigators and Research Physician: Design of the protocol, registration and conduct of the trial. Preparation of investigators brochure and case report forms. Organization of meetings of the steering committee Publication of study reports.

   - Lead Investigators: In each participating Primary Health Center, the principal investigator (Doctor of Family Medicine) will be identified, which will be responsible for the identification, patient information and recruitment.

   - Data manager: Data entry, analysis and maintenance of the computer system used.

   - Patient Security Committee: Within the team, a healthcare professional and an expert patient will control the development of the clinical trial, ensuring that is safe for the volunteers and that the project materializes as designed. A quarterly report will be issued reflecting a degree of compliance from 0 to 5 where 0 is the total absence of protocol compliance and 5 is absolute compliance. This commission will also be the communication vehicle between the volunteers and the research team for the resolution of doubts or attention to suggestions.

   - Management Committee: (Principal Investigators, Monitor, Medical Investigator, Administrator) Study planning, randomization, organization of meetings, provide annual development report and ethics committee.
10. DATA MONITORING

    10.1. Formal committee

    Although this trial focuses on a psychoeducational intervention, investigators will conduct quarterly reviews with the Patient Safety Committee and the Management Committee to assess patient feedback. If the information provided by the patients or the data analyzed at the time negatively affects the patients' clinic, the appropriate modifications are made or, in your case, the suspension.

    10.2. Intermediate analysis

    An interim analysis on the primary endpoint will be performed when 50% of participants have been randomized and completed the 6-month follow-up. An independent statistician, blinded for treatment allocation, will perform an interim analysis. The statistician will report to the Patient Safety Committee, which will decide on the continuation of the trial and will report to the central Ethics Committee.

    10.3. Auditing

    The clinical trial will have a monitor who will make visits to give support and solve problems. The monitor will:
    * discuss the protocol in detail and identify and clarify any areas of weakness
    * audit the quality and general integrity of the data
    * interview researchers and coordinators
    * confirm that the centre has complied with the protocol requirements
    * verify that all adverse events were documented in the correct format and that they are consistent with the protocol definition
    * Verify documentation: protocol and informed consent, the corresponding approvals, patient reports and documentation of dropouts and adverse events.

    The scheduling of follow-up visits will depend on patient enrollment, site status, and other commitments. Investigators must be available to meet with monitors.
11. ETHICAL ASPECTS

    11.1 Approval of research ethics

    The study design and subsequent development follow the recommendations for biomedical research in humans reflected in the Declaration of Helsinki through the World Medical Association. The patient will be informed verbally and with the delivery of a written document of the characteristics of the study, objectives, benefits and possible derived damages. Participation is voluntary and the patient will perform this right, contained in the Principle of Patient Autonomy, by signing the informed consent. This protocol and the Informed Consent have been reviewed and approved with applicable regulations in research and human subjects by the corresponding Ethics Committee (Virgen del Rocío University Hospital, Seville, Spain) with the code 1589-N-19 after modifying a correction suggested minor (update of the date of the Official Data Protection Law).

    11.2 Consent or assent

    Family Medicine specialists at the Public Primary Health Center will present the trial to patients and provide a background document explaining the study. Patients, after receiving verbal and written information, will have the opportunity to discuss or consult the information provided. The family doctor will get the signed informed consent of the patients who accept to participate in the trial. Information documents and consent forms are provided for all participants. The information document will be kept by the patient and the informed consent with the names, surnames and ID will be kept in a file with a unique password for each participating doctor. Once a week two of the researchers will collect the paper documents and take them to the Research Unit of the Hospital San Juan de Dios del Aljarafe, where the data will be coded and randomized once the identity of the patient is known. These documents will be protected in a closed filing cabinet belonging to the Head of the Investigation Unit.

    As it is a psychoeducational intervention versus no intervention, the patient's knowledge of the group to which has been assigned could condition the responses in the evaluation. To minimize biases secondary to knowledge of the assigned therapy, two information sheets have been designed. One of them describes in a general way what the study will consist of. This will be delivered to all participants recruited by primary care physicians. The second, in which the workshop is described in more detail, will be given only to patients who have been randomly included in the intervention group. It will be delivered at the beginning of the first workshop, being able to resolve any doubt in this regard. At this point, the patient can drop out of the study if they disagree.
12. CONFIDENTIALITY

For the safe handling of patient information:

1. The participants' medical record number will be coded and depersonalized, replacing the participant's identification information with an unrelated number.
2. The data and the link code will be stored in a separate database using encrypted digital files within password-protected folders and storage media to which only the statistical professional of the study who only participates in the analysis of the data will have access. data. The Management Committee will have access to the data to carry out audits, without knowing the link code of each patient and therefore the identity.
3. The confidentiality of the data will also be preserved when the data is transmitted over the Internet through the virtual private network of Hospital San Juan de Dios del Aljarafe.

The treatment, communication and transfer of personal data of all participating subjects will comply with the provisions of "Organic Law 3/2018, of December 5, Protection of Personal Data and Guarantee of Digital Rights". Following the aforementioned legislation, the patient can exercise the rights of access, modification, opposition and cancellation of the data, for which they must contact the Patient Safety Committee. The data collected for the study will be identified by a code and only a professional can relate this data to the patient and the medical history. Personal data will be used exclusively for scientific or statistical research purposes and will not be communicated or transferred to third parties, nor will they be subject to automated decisions or international transfers. Personal data, once they are no longer necessary, will be kept under the legally established deadlines, after which they will be deleted. Therefore, the identity of the patient will not be revealed to anyone, except for exceptions such as a medical emergency or a legal requirement. The processing of personal data will comply with the requirements described in the RGPD (General Data Protection Regulation).

If at any time the patient considers that the use of the data does not correspond to that described above, he or she may exercise the affected rights, in the terms provided by the regulations, as well as file a claim with the Control Authority Data Protection Agency ). In this sense, patients can go to Avenida. San Juan de Dios, s / n, CP 41930 Bormujos, Sevilla or contact our Data Protection Delegate through the email C15_DPO@sjd.es.

In compliance with article 12 of Law 14/2007 of July 3 on Biomedical Research, which establishes as principles and guarantees in this field of action the requirement of a favourable report issued by the Research Ethics Committee before the development of any project of research on human beings, this project and all the related material that was provided to the subject have been sent to the CEIC of the University Hospital Virgen del Rocío for evaluation and after the indicated corrections, the favourable opinion dated 23/10/2019 and the Internal Code of the project 1589-N-19 have been given.

As it is a non-pharmacological clinical trial, with a low level of intervention and no commercial purpose, according to sections 2 and 4 of article 9 of Royal Decree 1090/2015 on the regulations on methodology and regulation of clinical trials in Spain, contracting insurance would not be mandatory.

13. DECLARATION OF INTERESTS

The authors have no conflicts of interest to declare

ELIGIBILITY:
INCLUSION CRITERIA:

* People over the age of 18.
* People with mCNCP served for this reason in the Primary Care Centres depend on Hospital San Juan de Dios del Aljarafe, who follow regular specific treatment on the WHO analgesic scale and who have accepted, after information and informed consent signature, their participation in this study.
* Able to read and write Spanish.

EXCLUSION CRITERIA:

* Patients who have received interventional analgesic treatment in the year for the current disease.
* Have followed program or maintain out-of-hospital therapy similar to the one this study focuses on.
* Have had surgery or been on a waiting list during the study.
* Severe or decompensated systemic disease.
* Active cancer disease.
* Psychiatric pathology, epilepsy or cognitive impairment.
* Abuse drug addiction.
* Accidents or new Injuries that may increase the perception of pain during the study.
* Labor litigation due to pain.
* Language barrier.

LOSS CRITERIA:

* Voluntary abandonment of the study.
* Absence of one or more workshop sessions
* Partial or complete loss of telephone follow-up.
* Incomplete data collection.
* Exitus.
* Present any suspicious symptoms of COVID-19 disease collected by phone call the day before the workshop or communicate direct contact with a person infected in the previous days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain perception | Baseline and six months.
  It is measured by Verbal Numerical Rate Scale (NVRS). The NVRS will be used for its simplicity and reproducibility and in patients without cognitive impairment has a compliance close to 100%. Quantitative result by 0 to 10, where 0 is painless and 10 is as much pain as possible.
Change from Baseline Quality of life | Baseline and six months.
  It is measured by the EuroQol-5D questionnaire (EQ-5D). The EQ-5D is an instrument which evaluates the generic QoL with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit an index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status). We have used this questionnaire because its analysis of internal consistency shows high Cronbach coefficients.

SECONDARY OUTCOMES:
Gender. | Baseline.
  Dichotomous variable: "female" or "male".
Age. | Baseline.
  Quantitative variable: number of years of age.
Weight. | Baseline.
  Quantitative variable: number of kilograms in weight.
Height. | Baseline.
  Quantitative variable: number of centimeters in height. It is measured with a wall meter in the family medicien consult.
Body Mass Index (BMI). | Baseline.
  Quantitative variable: BMI will be expressed in: kilograms of weight/(height in meters)x2. It is calculated from the outcome 5 and 6.
% of patients with more than one type of pain in addition to mCNCP | Baseline.
  The number of participants who have one of the four possibilities of pain that can coexist with mCNCP. It is measured by a question with this options: "neuropathic", "visceral", "other", "none".
Pain evolution time. | Baseline.
  Quantitative variable: number of months with mCNCP until the start of the study.
Changes from Baseline analgesic pharmacological treatment defined by the WHO therapeutic scale at 6 months. | Baseline and six months.
  The incidence of changes in the type of analgesic drug treatment will be measured by one of the following nominal variables: "1= non-opioids +/- adjuvants"; "2= weak opioids +/- non-opioids +/- adjuvant"; "3= strong opioids +/- non-opioids +/- adjuvant".
Changes from Baseline amount of analgesic pharmacological treatment at 6 months. | Baseline and six months.
  The incidence of changes in the amount of analgesic drug treatment will be measured by one of the following nominal variables: "1= without requiring treatment"; "2= less treatment than 6 months ago"; "3= same treatment as 6 months ago"; "4= more treatment than 6 months ago".
Rate of smoking consumption. | Baseline.
  The rate of consumption will be calculated by choosing one of the following nominal variables: "1= never"; "2-=only in weekends and holidays"; "3= daily"; "4= I used to smoke but no longer".
Incidence of physical exercise practice. | Baseline.
  The incidence of the practice of physical exercise in specialized centres, home or outdoors by choosing one of the following nominal variables: "1- never", "2- less than one day a week", "3- 2 to 4 days a week", "4- 5 to 7 days a week".
Rate of alcohol consumption. | Baseline.
  The rate of consumption by choosing one of the following nominal variables: "1- never", "2- only in weekends and holidays", "3- daily", "4- used to drink but no longer".
% of patients with other concomitant chronic pathologies. | Baseline.
  Incidence of any type of disease with an evolution of more than six months that the participants present at the time of the evaluation by choosing one or more of the following items: "Depression"; "Anxiety"; "Insomnia", "Another mental illness"; "Cardiopulmonary disease"; "Cerebrovascular disease", "Chronic arterial disease", "Diabetes 1 and/or 2"; "Fibromyalgia"; "Celiac Disease"; "Inflammatory bowel disease", "Rheumatoid disease"; "Autoimmune disease"; "Disease of the nervous system"; "Thyroid disease", "Other", "None".
% of patients with family history of chronic pain. | Baseline.
  Number of patients with a family history of chronic pain during childhood. It is measured by choosing one of the following items: "Yes", "no", "don't know", "no answer".
Educational level. | Baseline.
  Level of studies before the start of the study by choosing one of the following items: "without studies", "primary education", "secondary education", "license", "diploma", "master", "doctorate", "degree", "other").
Habitual residence. | Baseline.
  Locality of the Aljarafe (Seville, Spain).
Marital status. | Baseline.
  Nominal variable: "Single", "married", "separated", "divorced", "widowed", "living together without marriage", "other").
Incidence of caregivers among participants. | Baseline.
  The number of participants with people who need their care daily (minors, the elderly or people with some type of disability) by answering:"Yes"; "No".
Employment situation. | Baseline.
  Nominal variable: "no employment but in active search", "no employment but no active search", "self-employed", "active without employment contract", "temporary work disability", "permanent work disability", "retired", "other".
Changes from Baseline Emotional Coping Strategies by the Reduced Chronic Pain Coping Questionnaire at 6 months. | Baseline and six months.
  The Reduced Chronic Pain Coping Questionnaire has shown validity equivalent to the non-reduced questionnaire, maintaining its internal consistency. In addition, in practice, it is a reliable, valid and easy-to-use instrument. With five possible answers ("never = 1", "rarely = 2", "neither many nor few = 3", "many times = 4", "always = 5") it is asked to define the frequency of use of one of the six coping strategies: religion, catharsis (search for socio-emotional support), distraction, mental self-control, self-affirmation and search for information (search for instrumental social support) distributed in 24 items in total. It gives us information about the adaptive strategy that has the most points in the assessment and that is predominant in each participant. The objective of this questionnaire is not to measure the degree of coping but to identify which adaptive strategies coexist with a better quality of life and lower perception of pain.
The rate of adherence to treatment. | Baseline, one, three and six months.
  The rate of adherence to treatment using the dichotomous answer "yes" (= 100% compliance with the treatment); "no" (=without 100% compliance with the treatment).
Incidence of causes of non-adherence to treatment. | Baseline, one, three and six months.
  The incidence of causes in the % of patients who have registered "non-adherence to treatment" using one of the following nominal variables: "forgotten", "refusal to take", "clinical improvement", "appearance of side effects", "other ".
Changes from Baseline Sleep Quality (Oviedo Questionnaire) at 6 months. | Baseline and six months.
  The Oviedo Questionnaire will be used for its simplicity and for a Cronbach's alpha coefficient for its internal consistency of 0.76 with adequate concurrent validity when compared with the Hamilton scale (Pearson's r of 0.78). With 15 items, 13 of them are grouped into 3 subscales: subjective satisfaction of sleep, insomnia and hypersomnia. The remaining 2 items provide information on the use of sleep aid or the presence of adverse phenomena during sleep. Each item is scored from 1 to 5, except for the subjective satisfaction of sleep that is made from 1 to 7. The subscale of insomnia ranges from 9 to 45, where a higher score equates to higher severity of insomnia.
Changes from Baseline Global Family Unit Operation (Family Apgar Test) at 6 months | Baseline and six months.
  The Family Apgar Test measures the global family unit operation, using five possible answers ("never"-1, "almost never"-2, "sometimes"-3, "almost always"-4, "always"-5) to seven questions you get an overall score that defines family functionality (normal 17-20, mild dysfunction 16-13, moderate dysfunction 12-10, severe dysfunction < 9). We have used this instrument for including friends in the perception of family dynamics, for its validity and reliability (Cronbach's alpha 0.84), whether it is self-completed or heteroadministered.
Changes in the frequentation of Medical Services during the study per patient. | Baseline, one, three and six months.
  Expressed in number of emergency consultations at home or in any health centre and the number of days of work disability caused by the intensification of pain. In addition to the direct questions to the patient, the data will be confirmed through the public health system database.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Sánchez Gutiérrez, MD, Principal Investigator — Hospital San Juan de Dios del Aljarafe (Seville, Spain); Adriana Rivera Sequeiros, Study Chair — Hospital San Juan de Dios del Aljarafe (Seville, Spain); Eugenia Gil García, Study Director — Schooll of Podiatry, Nursing and Physiotherapy. University of Seville. Spain; Jose Manuel López-Millán Infantes, MD, Study Director — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital San Juan de Dios del Aljarafe, Bormujos, Sevilla, Spain

IPD SHARING:
Plan to Share IPD: Yes
First, share the protocol and consent of the clinical trial through the ClinicalTrials.gov registry.
  Second, share the results of the study once it is finished, through congress and scientific journals.
Supporting Information: Study Protocol, ICF
Time Frame: Registration and consent will be available from the beginning of the study on ClinicalTrials.gov.
  The results will be published once the study is finished (2 years)
Access Criteria: ClinicalTrials.gov registry

REFERENCES:
- [Background] Hassed C. Mind-body therapies--use in chronic pain management. Aust Fam Physician. 2013 Mar;42(3):112-7. PMID 23529519
- [Background] Crofford LJ, Casey KL. Central modulation of pain perception. Rheum Dis Clin North Am. 1999 Feb;25(1):1-13. doi: 10.1016/s0889-857x(05)70052-1. PMID 10083956
- [Background] Kratz AL, F Murphy J 3rd, Kalpakjian CZ, Chen P. Medicate or Meditate? Greater Pain Acceptance is Related to Lower Pain Medication Use in Persons With Chronic Pain and Spinal Cord Injury. Clin J Pain. 2018 Apr;34(4):357-365. doi: 10.1097/AJP.0000000000000550. PMID 28877136
- [Background] Rethorn ZD, Pettitt RW, Dykstra E, Pettitt CD. Health and wellness coaching positively impacts individuals with chronic pain and pain-related interference. PLoS One. 2020 Jul 27;15(7):e0236734. doi: 10.1371/journal.pone.0236734. eCollection 2020. PMID 32716976
- [Background] Cherkin DC, Sherman KJ, Balderson BH, Cook AJ, Anderson ML, Hawkes RJ, Hansen KE, Turner JA. Effect of Mindfulness-Based Stress Reduction vs Cognitive Behavioral Therapy or Usual Care on Back Pain and Functional Limitations in Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA. 2016 Mar 22-29;315(12):1240-9. doi: 10.1001/jama.2016.2323. PMID 27002445
- [Background] Crofford LJ. Chronic Pain: Where the Body Meets the Brain. Trans Am Clin Climatol Assoc. 2015;126:167-83. PMID 26330672
- [Background] Theadom A, Cropley M, Smith HE, Feigin VL, McPherson K. Mind and body therapy for fibromyalgia. Cochrane Database Syst Rev. 2015 Apr 9;2015(4):CD001980. doi: 10.1002/14651858.CD001980.pub3. PMID 25856658
- [Background] Morone NE, Greco CM, Moore CG, Rollman BL, Lane B, Morrow LA, Glynn NW, Weiner DK. A Mind-Body Program for Older Adults With Chronic Low Back Pain: A Randomized Clinical Trial. JAMA Intern Med. 2016 Mar;176(3):329-37. doi: 10.1001/jamainternmed.2015.8033. PMID 26903081
- [Background] Stanos S. Focused review of interdisciplinary pain rehabilitation programs for chronic pain management. Curr Pain Headache Rep. 2012 Apr;16(2):147-52. doi: 10.1007/s11916-012-0252-4. PMID 22427179
- [Background] Anheyer D, Haller H, Barth J, Lauche R, Dobos G, Cramer H. Mindfulness-Based Stress Reduction for Treating Low Back Pain: A Systematic Review and Meta-analysis. Ann Intern Med. 2017 Jun 6;166(11):799-807. doi: 10.7326/M16-1997. Epub 2017 Apr 25. PMID 28437793
- [Background] Hilton L, Hempel S, Ewing BA, Apaydin E, Xenakis L, Newberry S, Colaiaco B, Maher AR, Shanman RM, Sorbero ME, Maglione MA. Mindfulness Meditation for Chronic Pain: Systematic Review and Meta-analysis. Ann Behav Med. 2017 Apr;51(2):199-213. doi: 10.1007/s12160-016-9844-2. PMID 27658913
- [Background] Malfliet A, Kregel J, Meeus M, Danneels L, Cagnie B, Roussel N, Nijs J. Patients With Chronic Spinal Pain Benefit From Pain Neuroscience Education Regardless the Self-Reported Signs of Central Sensitization: Secondary Analysis of a Randomized Controlled Multicenter Trial. PM R. 2018 Dec;10(12):1330-1343.e1. doi: 10.1016/j.pmrj.2018.04.010. Epub 2018 May 9. PMID 29753112
- [Background] Cuenda-Gago JD, Espejo-Antunez L. [Effectiveness of education based on neuroscience in the treatment of musculoskeletal chronic pain]. Rev Neurol. 2017 Jul 1;65(1):1-12. Spanish. PMID 28650061
- [Background] Louw A, Zimney K, Puentedura EJ, Diener I. The efficacy of pain neuroscience education on musculoskeletal pain: A systematic review of the literature. Physiother Theory Pract. 2016 Jul;32(5):332-55. doi: 10.1080/09593985.2016.1194646. Epub 2016 Jun 28. PMID 27351541
- [Background] Patel K, Sutherland H, Henshaw J, Taylor JR, Brown CA, Casson AJ, Trujillo-Barreton NJ, Jones AKP, Sivan M. Effects of neurofeedback in the management of chronic pain: A systematic review and meta-analysis of clinical trials. Eur J Pain. 2020 Sep;24(8):1440-1457. doi: 10.1002/ejp.1612. Epub 2020 Jun 30. PMID 32502283
- [Background] Gatchel RJ, McGeary DD, McGeary CA, Lippe B. Interdisciplinary chronic pain management: past, present, and future. Am Psychol. 2014 Feb-Mar;69(2):119-30. doi: 10.1037/a0035514. PMID 24547798
- [Background] Hassan S, Zheng Q, Rizzolo E, Tezcanli E, Bhardwaj S, Cooley K. Does Integrative Medicine Reduce Prescribed Opioid Use for Chronic Pain? A Systematic Literature Review. Pain Med. 2020 Apr 1;21(4):836-859. doi: 10.1093/pm/pnz291. PMID 31755962
- [Background] Pergolizzi JV Jr, Raffa RB, Rosenblatt MH. Opioid withdrawal symptoms, a consequence of chronic opioid use and opioid use disorder: Current understanding and approaches to management. J Clin Pharm Ther. 2020 Oct;45(5):892-903. doi: 10.1111/jcpt.13114. Epub 2020 Jan 27. PMID 31986228
- [Background] Henningfield JE, Ashworth JB, Gerlach KK, Simone B, Schnoll SH. The nexus of opioids, pain, and addiction: Challenges and solutions. Prev Med. 2019 Nov;128:105852. doi: 10.1016/j.ypmed.2019.105852. Epub 2019 Oct 18. PMID 31634511
- [Background] Gatchel RJ, Okifuji A. Evidence-based scientific data documenting the treatment and cost-effectiveness of comprehensive pain programs for chronic nonmalignant pain. J Pain. 2006 Nov;7(11):779-93. doi: 10.1016/j.jpain.2006.08.005. PMID 17074616
- [Background] Herman PM, Anderson ML, Sherman KJ, Balderson BH, Turner JA, Cherkin DC. Cost-effectiveness of Mindfulness-based Stress Reduction Versus Cognitive Behavioral Therapy or Usual Care Among Adults With Chronic Low Back Pain. Spine (Phila Pa 1976). 2017 Oct 15;42(20):1511-1520. doi: 10.1097/BRS.0000000000002344. PMID 28742756
- [Background] Palylyk-Colwell E, Wright MD. Tiered Care for Chronic Non-Malignant Pain: A Review of Clinical Effectiveness, Cost-Effectiveness, and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Feb 12. Available from http://www.ncbi.nlm.nih.gov/books/NBK543512/ PMID 31291071
- [Result] McCracken LM, Vowles KE, Eccleston C. Acceptance of chronic pain: component analysis and a revised assessment method. Pain. 2004 Jan;107(1-2):159-66. doi: 10.1016/j.pain.2003.10.012. PMID 14715402

DOCUMENTS (1):
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT04696107/ICF_000.pdf